CLINICAL TRIAL: NCT03229876
Title: A Safety and Efficacy Study of CD19-UCART (Allogeneic Engineered T-cells Expressing Anti-CD19 Chimeric Antigen Receptor) in Patients With Relapsed or Refractory B-cell Hematologic Malignancies
Brief Title: Safety and Efficacy Evaluation of CD19-UCART
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Bioray Laboratories (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Zhejiang University (Other); Second Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018CAR-00CH1
Record Dates: First submitted 2017-07-19; First posted 2017-07-26 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-03

CONDITIONS: Acute Lymphoblastic Leukemia (ALL); Non Hodgkin Lymphoma (NHL)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-UCART (Experimental): All patients will be treated with 1 injection of CD19-UCART. Three escalating dose-levels (1.0-2.0x10^6/kgBW, 2.5-5.0x10^6/kgBW, 5.5-10.0x10^6/kgBW) of CD19-UCART will be evaluated using a 3+3 design. Each CD19-UCART injection will be administered at Day 0.
  Interventions: Biological: CD19-UCART

INTERVENTIONS:
Biological: CD19-UCART — A conditioning therapy with cyclophosphamide and fludarabine will be conducted before CD19-UCART injection. VP16 can be added to the conditioning therapy.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ascending doses of CD19-UCART in patients with relapsed or refractory B-cell hematological malignancies.

DETAILED DESCRIPTION:
CD19-UCART is a kind of "off-the-shelf" product originated from health donor's PBMC.This is a open-label, dose estilation study to evaluate the safety and anti-tumor efficacy of CD19-UCART in the treatment of relapsed or refractory B-cell hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participating in this clinical study and signing the informed consent form; The estimated survival period is at least one month;
2. No other serious cardiopulmonary diseases, and normal liver and kidney functions (except for subjects with tumor lesions in their liver and kidneys);
3. Failure of T cell isolation during autologous CART preparation or failure of CART amplification or failure to complete apheresis or disease progression resulting in patients not benefiting from autologous CAR-T cell therapy; Or: T cell percentage in PBMC of peripheral blood ≤ 10%; Or the disease is not effectively controlled within one month after autologous CAR-T transfusion, and the patient cannot receive CAR-T transfusion again;
4. Flow cytometry within two months demonstrated positive expression of CD19 in the tumor (positive rate 50%-90%; Or biopsy ≥ 50% within 6 months; Or obtaining a biopsy again);
5. Hematological indicators: 1) WBC count ≥ 1.5× 10^9/L; Absolute value of neutrophils ≥ 0.8× 10^9/L; Lymphocyte count ≥0.1×10^9/L;2) Hemoglobin ≥ 60g/L;3) Platelet count ≥20×10^9/L;
6. Biochemical indicators (except for subjects with tumor foci in liver and kidney): Total bilirubin (TBIL)≤1.5 times the Upper Limits of Normal (ULN); AST and ALT≤1.5 *ULN; Scr and BUN)≤1.5*ULN; Biochemical indicators in subjects with liver and kidney invasion should meet: Total bilirubin (TBIL)≤5 *ULN;AST and ALT≤5*ULN; Scr and BUN ≤ 5*ULN;
7. Cardiac function: Good hemodynamic stability, and the left ventricular ejection fraction (LVEF) ≥ 55%;
8. Serum viral EBV-DNA, CMV-DNA, HIV antibody and syphilis antibody, HBV, HCV virus quantification were all negative;
9. ECOG activity status score: 0-2 points;
10. Female subjects must have access to effective contraceptive measures (e.g., oral prescription contraceptives, injectable contraceptives, intrauterine devices, double blocking, contraceptive patches, male partner sterilizations) throughout the study period; Serum or urine pregnancy test results must be negative at screening and throughout the study;
11. Willing to comply with the rules established in this protocol;
12. Patients with relapsed/refractory CD19-positive acute B-cell leukemia (B-ALL, with the age of 1-60 years) or relapsed/refractory B-cell non-Hodgkin's lymphoma (B-NHL, with the age of 5-65 years).

Exclusion Criteria:

1. Pregnant or lactating women;
2. The following drugs or treatments should be excluded:High-dose glucocorticoids were used within 72h prior to UCAR-T infusion, except for physiological alternative therapies;Allogeneic cell therapies such as donor lymphocyte transfusion within 6 weeks prior to UCAR-T transfusion;GVHD treatment;
3. Single extramedullary relapse B-ALL;
4. Suffering from severe mental disorder;
5. Active autoimmune diseases requiring immunotherapy;
6. History of other malignant tumors;
7. Patients with severe cardiovascular disease;
8. Organ function is in the following abnormalities;
9. Total bilirubin > 1.5 times the upper limit of normal unless the patient is Gilbert's syndrome;
10. Partial thromboplastin time or activated partial thromboplastin time or international normalized ratio >1.5*ULN；in the absence of anticoagulant therapy;
11. There is an active infectious disease or any major infectious event requiring high-level antibiotics;
12. Any condition that, in the opinion of the investigator, may increase the subject's risk or interfere with the test results.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) occurence | Baseline up to 35 days after T cell infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria

SECONDARY OUTCOMES:
Objective Response Rate | At 12 weeks, and overall
  The total response rate after 90 days of treatment with study drug (overall response rate for ALL= CR+CRi; for NHL=CR+PR);
Day 90 progression-free survival | Assessed up to 3 months
  The 90-day progression-free survival rate following drug therapy.

OTHER OUTCOMES:
UCART cell survival time | up to 1 year after infusion
  The number of UCART cells surviving in the body within 90 days after receiving the study drug;
Progrssion-free survival | up to 2 years after infusion
  The time from treatment with study drug to tumor progression or death.
Overall survival | up to 2 years after infusion
  the time from treatment with study drug to death by any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, Professor, Principal Investigator — First Affliated Hospital of Zhengzhou University; He Huang, Professor, Principal Investigator — First Affliated Hospital of Zhejiang University
Locations (2):
- China (2):
  - First Affliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - First Affliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No